CLINICAL TRIAL: NCT06445816
Title: Does the Level of Pain in Pediatric Oncology Patients Affect the Level of Psychological Resilience in Parents?
Status: Active, not recruiting | Type: Observational
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Bahar Nur Kanbur, Assistant Professor, Istanbul Gelisim University
Other Study IDs: Istanbul Gelişim Üniversity
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Pain; Pediatric Oncology; Psychological Resilience
MeSH Terms: conditions — Pain | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: chemotherapy — * Parents whose consent was obtained will be asked to fill out the Mother and Child Information Collection Form and Psychological Resilience Scale, respectively.
  * Immediately after receiving chemotherapy, the pain levels of the children will be measured with the Facial Expressions Pain Scale - Faces Pain Scale-Revised (FPS-R).
  * The psychological resilience scale will be applied to mothers.

SUMMARY:
Resilience is defined as generating coping strategies for the problems and situations that individuals face throughout their lives and developing these strategies in each new situation. While some individuals become helpless in the face of difficulties and give up the struggle, other individuals recover quickly in the face of difficulties and use coping methods well. Accordingly, these individuals have higher levels of crisis management and coping with stress.

DETAILED DESCRIPTION:
Psychological resilience is defined as the process of adaptation, the power of recovery or the ability to successfully overcome change/disasters against significant sources of stress such as a trauma, a threat, a tragedy or family and relational distress, serious health problems, workplace and financial problems. At the same time, psychological resilience, as a personality trait, is also used to mean the power to recover quickly, the power to overcome difficulties, resilience, flexibility and robustness. Individuals who are successful in repairing the psychological destruction that occurs as a result of negative emotional states are considered to be strong individuals in terms of psychological resilience.

Identification of protective factors Psychological resilience is a dynamic process resulting from the interaction of risk factors and protective factors. In the literature, the most frequently emphasized characteristics when defining psychological resilience are risk factors, protective factors that mitigate the impact of negative events and adaptation to risk factors.

Personal risk factors include anxious temperament, health problems, lack of self-confidence, inability to use effective coping mechanisms, inability to express oneself effectively, aggressive personality, pessimistic perspective.

Familial risk factors include lack of healthy family relationships, domestic violence, loss of parents, neglect and abuse in the family, and negative relationships.

Environmental risk factors include low socio-economic level, lack of positive role models, unemployment and migration.

Protective factors are situations that increase the individual's adaptation to all risk factors and improve the individual's competencies. In other words, they are factors that reduce or eliminate the negative effects of risk factors. In research, risk factors and protective factors are analyzed in three stages: individual, familial and environmental It is stated that individuals with high levels of psychological resilience have a higher level of control over their behaviors compared to other individuals, believe that they can achieve higher success as a result of their efforts, have better social competence and responsibilities, and are more successful in solving problems. When we look at other characteristics of individuals with high psychological resilience, it is stated that they have the power and resilience to influence the people around them and to take advantage of upsetting events and to achieve results. It has also been found that individuals with high levels of resilience have high levels of self-confidence and less anxiety. These individuals like to struggle and do not like to give up. Individuals with low levels of psychological resilience have poor self-control capacity, withdraw from the environment, do not participate in social life and show resistance to change. Individuals with good resilience prefer to struggle by questioning their lives.

ELIGIBILITY:
Inclusion Criteria:

* Children will be between 4-18 years old
* Communicable children and families
* The child will be hospitalized for inpatient treatment

Exclusion Criteria:

* Outpatients
* Terminal patients
* Children whose parents cannot be reached will be excluded from work

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will consist of children between the ages of 4-18 and their parents who are being treated at the Oncology Clinic of Altınbaş University Medical Park Bahçelievler Hospital in Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Psychological resilience scale | 2 day
  The pain level of the child receiving chemotherapy will reduce the psychological resilience of the mother. In the schematic evaluation, the scoring method is free for measuring psychological resilience as high or low.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sevinç, Principal Investigator — Arel University
Locations (1):
- Istanbul Gelisim University, Istanbul, Avcılar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No